CLINICAL TRIAL: NCT05526118
Title: Advanced HIV: Outcomes for Rapid ART
Acronym: AHORA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Valley AIDS Council (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: VAC-AHORA-1
Record Dates: First submitted 2022-07-25; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: HIV-1-infection
Keywords: rapid start; rapid art initiation; bictegravir; hispanic; latinx; latinos; advanced HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AHORA group: All 50 prospective subjects are enrolled into a single cohort, all subjects must meet inclusion/exclusion criteria
  Interventions: Drug: Bictegravir/emtricitabine/tenofovir alafenamide

INTERVENTIONS:
Drug: Bictegravir/emtricitabine/tenofovir alafenamide — Patients who are ART-naive adults,18 years of age and older, diagnosed with HIV within 7 days of study entry who have a clinical (diagnosed Opportunistic Infection/AIDS-defining illness) or laboratory (CD4<200) diagnosis of advanced HIV, who are clinically appropriate for Rapid ART initiation, and are initiated on bic/f/taf per DHHS guidelines at their initial clinic visit will be monitored for time to viral suppression, efficacy and CD4 cell recovery over the course of 48 weeks.
  Other Names: Biktarvy

SUMMARY:
AHORA is designed as a single-arm, open label, non-comparative, real-world prospective, observational study evaluating the outcomes for viral control and CD4 recovery/immune reconstitution in predominantly Hispanic/Latinx patients of the Rio Grande Valley (RGV) with advanced HIV who are rapidly initiated on bictegravir/emtricitabine/tenofovir alafenamide (Biktarvy) at Valley AIDS Council (VAC) dba Westbrook Clinic (WBC). This research will help to fill data gaps still present for Biktarvy in a rapid start setting among an Hispanic/Latinx population, including those with advanced HIV.

DETAILED DESCRIPTION:
VAC is the primary provider of HIV prevention, education and testing services and the only Ryan White funded agency providing medical care and supportive services for people with HIV in the RGV. VAC provides services to over 1700 patients with HIV, 52% of patients at VAC are diagnosed with advanced HIV disease. Generally speaking, HIV clinical trials have often lacked representation and enrollment of patients of Hispanic/Latinx ethnicity, and those with advanced HIV and this study has the potential to fill in those data gaps.

For AHORA, data from ART-naive, newly diagnosed HIV-1+ adults (18 years of age and older) with late presentation (CD4<200 or diagnosed Opportunistic infection/AIDS-defining illness) initiated on Biktarvy within 7 days from diagnosis will be collected and analyzed. Patients will be enrolled through VAC's linkage to care and RAPIDO (Rapid Start) programs. Patients appropriate for Rapid ART initiation with Biktarvy will be recruited, with a goal of 50 enrollees. Patients who agree to participate will have data collected at weeks 1,4,12, 24, 36, and 48 weeks for evaluation of time to viral suppression and efficacy, as well as evaluation of CD4 cell recovery.

ELIGIBILITY:
Inclusion Criteria:

* ART-naive adults,18 years of age and older
* diagnosed with HIV within 7 days of study entry
* diagnosis of Advanced HIV: clinical (diagnosed Opportunistic Infection/AIDS-defining illness) or laboratory (CD4<200) diagnosis of advanced HIV.

Exclusion Criteria:

* Known severe renal impairment (CrCl <30 mL/min/1.73 m2);
* Known or suspected severe hepatic impairment or unstable liver disease (Child Pugh Class C);
* Use of rifamycins for treatment of OIs
* use of concomitant medications that would be contraindicated for coadministration with Biktarvy;
* OI diagnosis requiring initiation of OI treatment for >7 days prior to initiation of ART.
* pregnant at time of diagnosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced HIV in the Rio Grande Valley (RGV) of Texas who are receiving treatment services with Valley AIDS Council (VAC) dba Westbrook Clinic (WBC). 92% of patients receiving services at VAC/WBC identify as Hispanic/Latinx.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Viral Suppression | 24 weeks
  To evaluate efficacy and time to HIV viral suppression of Biktarvy in Rapid Start setting for persons with Advanced HIV

SECONDARY OUTCOMES:
Viral Suppression | 48 weeks
  To evaluate efficacy, continued viral suppression of Biktarvy through 48 weeks.
CD4 cell recovery | 48 weeks
  Secondary objectives would be to evaluate immune function recovery via absolute CD4 cell count
CD4 cell recovery | 48 weeks
  Secondary objectives would be to evaluate immune function recovery via percent CD4 cell count
CD4 cell recovery | 48 weeks
  Secondary objectives would be to evaluate immune function recovery via CD4/CD8 ratio

OTHER OUTCOMES:
post-hoc analyses to evaluate potential associations of baseline characteristics on viral suppression | 48-72 weeks
  Descriptive analysis will evaluate potential associations of baseline characteristics on primary endpoint outcomes/ HIV viral suppression: sex at birth
post-hoc analyses to evaluate potential associations of baseline characteristics on viral suppression | 48-72 weeks
  Descriptive analysis will evaluate potential associations of baseline characteristics on primary endpoint outcomes/ HIV viral suppression: age at HIV diagnosis
post-hoc analyses to evaluate potential associations of baseline characteristics on viral suppression | 48-72 weeks
  Descriptive analysis will evaluate potential associations of baseline characteristics on primary endpoint outcomes/ HIV viral suppression: CD4 nadir
Post-hoc analyses to evaluate potential associations of baseline characteristics on viral suppression | 48-72 weeks
  Descriptive analysis will evaluate potential associations of baseline characteristics on primary endpoint outcomes/ HIV viral suppression: initial HIV viral load
Post-hoc analyses to evaluate potential associations of baseline characteristics on viral | 48-72 weeks
  Descriptive analysis will evaluate potential associations of baseline characteristics on primary endpoint outcomes/ HIV viral suppression: patient reported treatment adherence
Post-hoc analyses to evaluate potential associations of baseline characteristics on viral | 48-72 weeks
  Descriptive analysis will evaluate potential associations of baseline characteristics on primary endpoint outcomes/ HIV viral suppression: medical insurance status
Post-hoc analyses to evaluate potential associations of baseline characteristics on viral | 48-72 weeks
  Descriptive analysis will evaluate potential associations of baseline characteristics on primary endpoint outcomes/ HIV viral suppression: housing status
Post-hoc analyses to evaluate potential associations of baseline characteristics on viral | 48-72 weeks
  Descriptive analysis will evaluate potential associations of baseline characteristics on primary endpoint outcomes/ HIV viral suppression: federal poverty level

IPD SHARING:
Plan to Share IPD: No
Coded data will be kept by sponsor for potential future use if patient subject consents to their data being used for future research. Presently there is no plan to share IPD. However, data obtained through this study may be provided to qualified researchers with academic interest in HIV. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party. Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).